CLINICAL TRIAL: NCT01760850
Title: Investigating a Breast and Cervical Cancer Intervention for Latinas in Western New York
Brief Title: Breast and Cervical Cancer Educational Intervention for Latinas in Western New York
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 105707; NCI-2012-02850 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Esperanza y Vida) (Experimental): Participants engage in the Esperanza y Vida educational information session for breast and cervical cancer.
  Interventions: Other: educational intervention; Other: questionnaire administration
- Arm II (control) (Active Comparator): Participants engage in an educational information session for diabetes.
  Interventions: Other: educational intervention; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Engage in the Esperanza y Vida educational information session for breast and cervical cancer
  Other Names: intervention, educational
  Arms: Arm I (Esperanza y Vida)
Other: educational intervention — Engage in an educational information session for diabetes
  Other Names: intervention, educational
  Arms: Arm II (control)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies a breast and cervical cancer educational intervention for Latinas in Western New York. An outreach program may help minority cancer patients overcome problems that keep them from receiving cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the extent of linguistic and cultural tailoring necessary to adapt Esperanza y Vida outreach programs for Hispanics in Western New York.

II. Evaluate the effectiveness of the Esperanza y Vida program intervention to increase breast and cervical cancer knowledge and screening behaviors in Hispanic participants compared to a control health education program on diabetes.

III. Determine the factors associated with and/or predictive of screening of Hispanics in Western New York (WNY) as compared to New York City (NYC) and Arkansas to describe how the intervention impacts barriers and motivations for screening in diverse Hispanic populations.

OUTLINE:

Key informant interviews with local "gatekeepers" of Hispanic culture groups in WNY and focus groups with Hispanic cancer survivors with screened and unscreened participants are conducted during the first phase of research. Participants are then randomized to 1 of 2 arms.

ARM I: Participants engage in the Esperanza y Vida educational information session for breast and cervical cancer.

ARM II: Participants engage in an educational information session for diabetes.

After completion of study treatment, participants are followed up at 2 and 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are generally healthy, ambulatory, and able to participate in social events in their communities
* No women, men, or children of any ethnic or social background are ever excluded from the educational programs, although recruitment will focus on Hispanic/Latinos
* Children may be present with parents, but will not be included in any research activities, unless they are emancipated minors (under 18 and married)
* Men are included in all of the research activities, but will not be included in the follow-up telephone surveys to assess breast and cervical screening as they do not obtain screening Pap smears, clinical breast exams, or mammograms; men may be asked about their intent to assist women in obtaining screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2015-04

PRIMARY OUTCOMES:
Screening rates | 2 months
  Intervention-group screening rates will be compared for evidence of increase over control-group screening rates using the Chi-square test, conducted as a one-sided test at alpha = 0.05. And in stratified analysis, screening rates across both states will be compared for evidence of an overall increase with intervention using the Cochran-mantel-Haenszel (CMH) test, conducted as a one-sided test at alpha = 0.05.
Screening rates | 8 months
  Intervention-group screening rates will be compared for evidence of increase over control-group screening rates using the Chi-square test, conducted as a one-sided test at alpha = 0.05. And in stratified analysis, screening rates across both states will be compared for evidence of an overall increase with intervention using the CMH test, conducted as a one-sided test at alpha = 0.05.
Knowledge acquisition | 2 months
  Knowledge acquisition within the intervention group will be assessed using the 1-sided paired t-test at alpha = 0.05, while differences in knowledge acquisition between groups will be assessed using Analysis of Covariance (ANCOVA).
Knowledge acquisition | 8 months
  Knowledge acquisition within the intervention group will be assessed using the 1-sided paired t-test at alpha = 0.05, while differences in knowledge acquisition between groups will be assessed using ANCOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Erwin, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States